CLINICAL TRIAL: NCT00024297
Title: A Multicenter Prospective Randomized Controlled Trial of Thrombosis Prophylaxis With Warfarin in Cancer Patients With Central Venous Catheters
Brief Title: Warfarin in Preventing Blood Clots in Cancer Patients With Central Venous Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research Campaign Clinical Trials Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CRC-WARP; CDR0000068909 (Registry Identifier: PDQ (Physician Data Query)); EU-20049; ISRCTN50312145 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register))
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2002-12

CONDITIONS: Thromboembolism
Keywords: thromboembolism
MeSH Terms: conditions — Thromboembolism | interventions — Warfarin

INTERVENTIONS:
Drug: warfarin

SUMMARY:
RATIONALE: Warfarin may be effective in preventing the formation of blood clots in patients with central venous catheters.

PURPOSE: Randomized clinical trial to study the effectiveness of warfarin in preventing blood clots in cancer patients who have central venous catheters.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the utility of warfarin in reducing thrombosis rates in cancer patients with central venous catheters.
* Compare the thrombosis rates in patients treated with different warfarin dosing schedules.
* Compare the adverse events and survival of patients receiving or not receiving this drug.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to sclerosant potential of cytotoxic regimen (low vs high), site of placement of catheter (peripheral vs central), and duration of drug administration (brief infusion (under 24 hours) vs prolonged infusion (24 hours and over)). Patients are randomized to 1 of 3 arms.

* Arm I: Patients receive no warfarin.
* Arm II: Patients receive oral warfarin daily beginning 3 days before placement of central venous catheter (CVC) and continuing until CVC is removed or thrombosis occurs.
* Arm III: Patients receive oral warfarin as in arm II, with dose adjustment after CVC placement to achieve and maintain INR level.

Patients are followed at 12 months.

PROJECTED ACCRUAL: A total of 1,400 patients (400 in arm I, 700 in arm II, and 300 in arm III) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cancer
* Planned placement of central venous catheter (CVC) for administration of chemotherapy

  * No use of CVC for additional purposes except for antibiotic therapy or blood products

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 2,000/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10 g/dL
* No congenital bleeding disorders

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No contraindication to warfarin
* No anatomic lesions that bleed (e.g., duodenal ulcers)
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior enrollment on this study
* No concurrent therapy that would interfere with study drug
* No concurrent warfarin

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Young, Study Chair — University Hospital Birmingham
Locations (38):
- United Kingdom (38):
  - Queen Elizabeth Hospital at University of Birmingham, Birmingham, England
  - City Hospital - Birmingham, Birmingham, England
  - Birmingham Heartlands and Solihull NHS Trust -Teaching, Birmingham, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Diana Princess of Wales Hospital, Grimsby, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Princess Royal Hospital, Hull, England
  - Ipswich Hospital NHS Trust, Ipswich, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Guy's and St. Thomas' Hospitals NHS Foundation Trust, London, England
  - St. George's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - South Tees Hospitals NHS Trust, Middlesbrough, Cleveland, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Royal Preston Hospital, Preston, England
  - Oldchurch Hospital, Romford, England
  - Royal South Hants Hospital, Southampton, England
  - Sandwell General Hospital, West Bromwich, England
  - Good Hope Hospital Trust, West Midlands, England
  - Airedale General Hospital, West Yorkshire, England
  - Royal Hampshire County Hospital, Winchester, England
  - New Cross Hospital, Wolverhampton, England
  - Worcester Royal Hospital, Worcester, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - Singleton Hospital, Swansea, Wales
  - Plymouth Hospitals NHS Trust, Plymouth